CLINICAL TRIAL: NCT04510181
Title: Effect of an Orally Administered Amino Acid-Based Blend on Human Growth Hormone (hGH) Levels and Fibromyalgia (FM) Symptoms: A Prospective, Open-Label, Single-Arm, Observational 24-Week Study in Adults With Poorly Controlled FM and Low hGH
Brief Title: Effect of an Amino-Acid-Based Blend on Human Growth Hormone (hGH) and Fibromyalgia (FM) Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pekarovics, Susan, MD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SePe-03-2020
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amino acid-based blend (Experimental): The amino acid-based blend will be administered PO daily for the study duration
  Interventions: Dietary Supplement: amino acid-based blend

INTERVENTIONS:
Dietary Supplement: amino acid-based blend — blended (listed in descending order) L-lysine, L-arginine, oxo-proline, N-acetyl-l-cysteine, L-glutamine, and Schizonepeta tenuifolia

SUMMARY:
The purpose of the study is to investigate the effect of the amino acid-based blend on growth hormone levels (measured by IGF-1) and clinical symptoms in individuals with treatment-resistant FM and low-normal hGH.

DETAILED DESCRIPTION:
Low hGH levels have been observed in approximately 1/3 of individuals with FM. Low hGH levels are hypothesized to contribute to inadequate treatment outcomes in many individuals with FM and several studies have demonstrated symptom improvement in individuals with FM and low hGH who received rhGH therapy. The amino acid-based blend represents a novel mechanism for increasing endogenous hGH production. It has been shown to produce an increase in endogenous hGH levels in healthy individuals by attenuating the inhibitory effect of somatostatin on hGH release. The amino acid-based blend may be a safe and effective treatment for FM in individuals with poorly controlled FM and low-normal hGH.

This study will investigate the effect of taking the amino acid blend on IGF-1 levels (a surrogate marker of the body's growth hormone levels), fibromyalgia symptoms, stress symptoms, body weight, and other cardiometabolic biomarkers in individuals with treatment-resistant FM and low-normal hGH.

After being informed about the study and potential risks, all eligible participants giving written informed consent will administer the amino acid-based blend daily. Standard care for fibromyalgia will continue.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of FM for at least 10 years, poorly controlled FM symptom, and receiving standard of care treatment at the Private Medical Practice of Susan Pekarovics, MD
2. Have low to normal levels of hGH (screening IGF-1 levels between the 15th and 50th percentile for age-appropriate levels)
3. Female participants of childbearing potential will agree to avoid pregnancy during the study.
4. Capable of giving signed informed consent

Exclusion Criteria:

1. Human growth hormone deficiency (GHD)
2. Individuals with a total score of ≥15 (indicating the presence of moderately severe major depression) or a score of >0 on Item 9 (suicidal ideation) on the Patient Health Questionnaire-9 (PHQ-9)
3. Pregnant women or women who wish to become pregnant
4. History of substance abuse
5. Previous treatment with recombinant human growth hormone (rhGH)
6. Individuals belonging to the following vulnerable populations: people with disabilities, people who cannot read, educationally disadvantaged, individuals with a serious or life threatening illness, prisoners, non-English speakers, economically disadvantaged individuals, employees of the study sponsor/site.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in IGF-1 | 24 weeks, 52 weeks
  change from baseline in IGF-1, a surrogate marker of hGH

SECONDARY OUTCOMES:
Fibromyalgia symptoms | 24 weeks, 52 weeks
  Change from baseline in score on the Revised Fibromyalgia Impact Questionnaire (FIQR, a 21-item self-report measure that estimates the severity and impact of FM. Score ranges from 0-100 with higher scores indicating greater severity/impact of FM)
Stress symptoms | 24 weeks, 52 weeks
  Change from baseline in score of the Perceived Stress Scale (PSS, a 10-item self-report measure that assesses the perception of stress. Total score ranges from 0-40 with higher scores indicating greater perceived stress)
Insulin-like growth factor binding protein-3 (IGFBP-3), an indicator of IGF-1 bioavailability | 24 weeks, 52 weeks
  Change from baseline
body weight (kg) | 24 weeks, 52 weeks
  Change from baseline
body mass index (BMI) | 24 weeks, 52 weeks
  Change from baseline
Blood pressure (systolic and diastolic) | 24 weeks, 52 weeks
  Change from baseline
HbA1c | 24 weeks, 52 weeks
  Change from baseline
Fasting total cholesterol | 24 weeks, 52 weeks
  Change from baseline
Fasting HDL cholesterol | 24 weeks, 52 weeks
  Change from baseline
Fasting LDL cholesterol | 24 weeks, 52 weeks
  Change from baseline
Fasting triglycerides | 24 weeks, 52 weeks
  Change from baseline
Fasting glucose | 24 weeks, 52 weeks
  Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Susan Pekarovics, MD, Principal Investigator — Pekarovics, Susan, MD
Locations (1):
- Private Medical Practics of Susan Pekarovics, MD, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset of selected variables that underlie results in a publication. Some data may not be amenable to complete anonymization and will not be shared to ensure appropriate confidentiality of participant's data.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after publication
Access Criteria: Upon appropriate data request by other scientists